CLINICAL TRIAL: NCT06512298
Title: Plasticizer Exposure and Its Consequences on Health
Acronym: PEACH
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Lukas Wisgrill, Principal Investigator, MD, Medical University of Vienna
Other Study IDs: 1716/2023; 10.55776/KLP1811624 (Other Grant/Funding Number: FWF)
Record Dates: First submitted 2024-07-06; First posted 2024-07-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Beta-thalassemia; Glioma; Healthy Controls; Transfusion-dependent Beta-Thalassemia; Intracranial Hemorrhages; Toxicity
Keywords: Plasticizer; Transfusion; Systems Biology; Immunology; Microbiome; Neuropharmacology; Pharmacokinetics; Pharmacodynamics; Exposomics
MeSH Terms: conditions — beta-Thalassemia; Glioma; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All collected samples will be analyzed for study purposes only. After completion of the study, left material will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Transfusion-dependent thalassemia major (TDTM): Patients suffering from homozygous transfusion-dependent Thalassemia Major.
- Thalassemia Minor: Patients suffering from heterozygous transfusion-independent Thalassemia Minor.
- Healthy controls: Healthy adult controls without any prevalent substance use (nicotine, alcohol etc.).
- Glioma patients: Adults with high/low-grade glioma, a tumor size > 3cm that require resection with access to the ventricular system without ventricular hemorrhage.
- ICU patients: Adults with brain hemorrhage (intracranial, subdural, subarachnoidal), treated with a ventricular shunt.
- Patients undergoing diagnostic lumbar-puncture (plastic-naive): Adults that receive a diagnostic lumbar puncture in an outpatient setting.

SUMMARY:
Plasticizers are chemicals commonly found in many everyday items, from food packaging to medical equipment. Although they are pervasive in our daily lives, researchers still don't have a clear picture of their long-term effects on human health. Evidence suggests that these substances might disrupt various biological functions such as the immune system, the balance of gut bacteria, hormone regulation, and brain processes. While some studies have linked plasticizer exposure to health issues, definitive data from human studies are still lacking.

The PEACH study aims to bridge these knowledge gaps by investigating how plasticizers affect human health. The study focuses on understanding how these chemicals are absorbed, distributed, and accumulated in the body across different groups of patients. The investigators are particularly interested in how plasticizers influence gut microbiota and the functionality of immune cells, as well as their effects on neurotransmitters involved in brain function.

A combination of patient data, systems biology, and laboratory models will be used to thoroughly assess the biological impacts of plasticizers. Advanced techniques such as mass spectrometry will aid in studying toxicokinetic properties, sequencing technologies will be used to examine immune effects, and radiouptake assays will be employed to explore interactions with neurotransmitter transport. This comprehensive methodology will provide new insights into the effects of both short-term and long-term exposure to plasticizers.

The PEACH study introduces innovative methods to the field, aiming to create a robust model for understanding how plasticizer compounds behave in the human body. It employs state-of-the-art techniques to assess the dynamics of these chemicals, marking a significant advancement in environmental health research.

DETAILED DESCRIPTION:
Wider research context: Industrial plasticizers are ubiquitous in modern society, utilized in products ranging from food packaging to medical supplies. Despite their widespread use, the health implications of chronic plasticizer exposure in humans remain inadequately understood. These substances potentially interfere and disrupt various biological processes, including immune activity, gut microbiota balance, endocrinological function, and neurophysiological health. Current epidemiological or exposure studies were able to pinpoint clinical associations with plasticizer exposures, but conclusive mechanistic human in vivo data are missing.

Research questions: The PEACH study is designed to fill critical gaps in the understanding of the biological implications of plasticizer exposure. The investigators aim to analyse the pharmacokinetics of plasticizers in different patient cohorts and elucidate their bioaccumulation, distribution, and metabolism. Thereby, the interplay between plasticizer exposure and metabolism, gut microbiota composition and immune cell functionality will be explored. Furthermore, the impact of plasticizer exposure on neurotransmitter physiology will be elucidated.

Approach: The study employs a comprehensive methodology that integrates the findings from clinical cohorts, systems biology approaches, and in vitro models. Three distinct work packages will examine pharmacokinetic properties via mass spectrometry, study immunological effects through advanced sequencing technologies & phenotypization, and investigate pharmacodynamic interactions with neurotransmitter transporters using human in-vitro assays. Longitudinal sampling from acute and chronic exposure cohorts will offer an evolving perspective on effects of plasticizer exposure.

Level of originality: The PEACH study introduces groundbreaking methodologies and scope to the investigation of plasticizer exposure. It aims to support the scientific community with first human in-vivo pharmacokinetic models for these compounds while utilizing high-throughput techniques for pharmacodynamic assessment, marking a notable advancement in the field.

ELIGIBILITY:
TDTM:

* Inclusion: Adult, homozygous ß-Thalassemia Major, transfusion dependency.
* Exclusion: Plastic implants, chronic infectious disease, pregnancy.

Thalassemia Intermedia/Minor:

* Inclusion: Adult, homozygous/heterozygous ß-Thalassemia Intermedia/Minor
* Exclusion: Plastic implants, chronic infectious disease, pregnancy, transfusion dependency

Healthy adults:

* Inclusion: Adult
* Exclusion: Chronic disease, plastic implants, infectious disease, pregnancy, anemia, medication-, drug-, or alcohol-abuse

Glioma patients:

* Inclusion: Adult, high/low-grade glioma, tumor larger then 3cm, resection with access to the ventricular system
* Exclusion: Large intraventricular hemorrhage, plastic implants, infectious disease

ICU patients:

* Inclusion: Adult, brain hemorrhage, external CSF drain from ventricle
* Exclusion: intraventricular hemorrhage, plastic implants, ECMO, hemodialysis, infectious disease

Patients undergoing diagnostic lumbar-puncture:

* Inclusion: Adult, diagnostic CSF sampling, outpatient setting
* Exclusion: Ventricular hemorrhage, plastic implants, infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two study cohorts will be recruited, one to study chronic exposure to plasticizers and another to analyze the "acute" penetration of plasticizers into the central nervous system. In total, 20 TDTM patients, 20 non-transfusion-dependent ß-thalassemia intermedia/minor patients, and 20 healthy controls will be recruited to study chronic exposure. To study the pharmacokinetics of acute transfusion-related accumulation of plasticizers within the CNS, 20 patients undergoing glioma resection, 20 ICU patients suffering from brain hemorrhage without ventricular collapse, and CSF from a cohort of medical-plastic-naïve patients undergoing diagnostic lumbar puncture in the outpatient setting (n=20) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Accumulation of plasticizers in transfused patients | 3 years
  Plasticizer concentrations (mmol/L) will be measured from the plasma of thalassemia major patients two weeks after the last pRBC-transfusion and compared to plasma levels of healthy controls of beta-thalassemia intermedia/minor patient using MANCOVA. Age, sex and liver/kidney retention will be taken into account as covariates and Tukey HSD or Scheffe tests used for even and uneven group sizes, respectively.

OTHER OUTCOMES:
Accumulation of plasticizers during storage in pRBC-bags | 1 year
  Biweekly measurements of blood-bag aliquots will be conducted, and concentrations of > 30 plasticizer analyzed. 15 of these (main compounds) will be used and subjected to repeated measures ANOVA with within group comparisons. The Sidak correction will be used as a post-hoc test.
Plasticizer release into the CSF of ICU-patients | 3 years
  The accumulation/release of plasticizers within/into the CSF (mmol/L) will be monitored longitudinally in relation to time (h) using repeated-measures ANCOVA with Sidak correction. Age, sex, as well as liver and kidney function will be considered as covariates.
Studying the accumulation of plasticizers within the CSF using a cross-sectional design | 3 years
  Accumulation of plasticizers within CSF will be analyzed using MANCOVA, taking age, sex, liver/kidney function as covariates. Thereby, abundancy (mmol/L) of plasticizers within the CNS will be compared between groups.
Pharmacodynamic analyses (IC50) | 3 years
  IC50 (mmol/L) values for neurotransmitter transport at SLC6 transporters will be derived upon co-incubation with plasticizers during the uptake of the transporters cognat substrate to describe the pharmacological profile of plasticizers and their interaction with neurotransmitter transport.
Pharmacodynamic analyses (Vmax) | 3 years
  Vmax values for neurotransmitter transport at SLC6 transporters (pmol/min) will be derived upon co-incubation with plasticizers during the uptake of the transporters cognat substrate to describe the pharmacological profile of plasticizers and their interaction with neurotransmitter transport.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No